CLINICAL TRIAL: NCT04951375
Title: Clinical Results of Arthroscopic Repair for Massive Rotator Cuff Tears of 14 Cases
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018054
Record Dates: First submitted 2021-06-17; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Rotator Cuff Tears
Keywords: Shoulder joint; Arthroscopy; Massive rotator cuff tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: arthroscopic repair — arthroscopic repair

SUMMARY:
This study retrospectively analyzed data of 14 cases of massive rotator cuff tears who were treated with arthroscopic repair by the same doctor from October 2015 to December 2017, aiming to explore the surgical methods and clinical effects of arthroscopic repair for massive rotator cuff tears.

DETAILED DESCRIPTION:
The preoperative and intraoperative data and patient information of 14 cases of arthroscopic repair of huge rotator cuff tears performed by Deputy Chief Physician Yang Yuping of the Institute of Sports Medicine of Peking University Third Hospital from January 2016 to August 2017 sort out. Collect and organize follow-up data on the recovery and motor function of patients 6 months after surgery and the latest follow-up (February 4 to March 3, 2018). Discuss the operation method, and statistically analyze the short-term curative effect of patients undergoing the operation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as massive rotator cuff tears and treated with arthroscopic repair from October, 2015 to December, 2017

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From October, 2015 to December, 2017, 14 cases of massive rotator cuff tears who were treated with arthroscopic repair by the same doctor were included.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
VAS | 6 months after surgery
  Pain visual analog scale
DASH | 6 months after surgery
  Arm, shoulder and hand dysfunction score
OSS | 6 months after surgery
  Oxford University Shoulder Score

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Yang, Study Director — Peking University Third Hospital
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No